CLINICAL TRIAL: NCT01295840
Title: QUARTET LEAD AND RESYNCHRONIZATION THERAPY OPTIONS To Investigate the Stimulatory Possibilities Offered by the Different Configurations Available for the Quartet Lead and Their Effect on Haemodynamic and Clinical Response.
Brief Title: Quartet Lead and Resynchronization Therapy Options
Acronym: QUARTO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CR 10-046-SP-HF
Record Dates: First submitted 2011-02-03; First posted 2011-02-15 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CRT therapy (No Intervention): Cardiac Resynchronization Therapy Defibrillator (CRT-D)
  Interventions: Device: Cardiac Resynchronization Therapy Defibrillator

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy Defibrillator — Cardiac Resynchronization Therapy Defibrillator
  Other Names: Promote Q. Model; Promote Quadra™.; Quartet®: Tetrapolar left ventricular lead. Model 1458Q.

SUMMARY:
The purpose of this Clinical Trial is to determine the percentage of patients whose hemodynamic response improves with the different configurations offered by the new Quartet® left ventricular lead, as a result of its four electrodes, with respect to the configurations offered by a standard bipolar lead.

Furthermore, the optimal stimulation configuration will be determined from a comparison with traditional configurations.

DETAILED DESCRIPTION:
This is a prospective, non-randomised, multi-centre, national, interventional clinical trial of a medical device.

This trial involves two visits: one at the beginning of the study, which will be undertaken in the seven days following implant, and another visit at 6 months after enrollment. It is recommended that the enrollment visit is undertaken as soon as possible after implantation, although the time window allows the timing to be adapted to each centre's standard practice. Resynchronization therapy in those patients suitable for participation in this trial is expected to begin once this enrollment visit has been completed.

Once data collection at enrollment visit has been completed, final device programming will be based on each investigator's criteria and will be undertaken following the standard practice of each centre.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a Cardiac resynchronization Therapy Defibrillator device (CRT-D) and a Quartet® quadripolar electrode from St Jude Medical (used in "Single Site Pacing" mode) implanted in the left ventricle.
2. Patients who have provided written informed consent
3. Patients who are in sinus rhythm.
4. Patients older than 18 years of age.

Exclusion Criteria:

1. Patients in atrial fibrillation at the time of the echocardiographic study of the enrollment visit.
2. Patients with valvular disease.
3. Patients in functional class New York Heart Association (NYHA) IV
4. Patients for whom echocardiography images suitable for determining the cardiac output cannot be obtained.
5. Patients whose device has been changed/upgraded.
6. Pregnant patients.
7. Patients who do not fulfill all the inclusion criteria.
8. Patients who are unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Francisco Javier Alzueta Rodríguez, PhD, Principal Investigator — Hospital Clínico Universitario Virgen de la Victoria
Locations (1):
- Hospital Clínico Universitario Virgen de la Victoria, Málaga, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment target is approximately 50 patients. Recruitment will be competitive, and will last for approximately 12 months, plus six months of follow-up. The trial will finish once all the patients have completed the follow-up.
Groups:
- No Arms: All patient have a Quartet Left Ventricular (LV) lead. No arms.
Period: Overall Study
Arm/Group | No Arms
Started | 51
Completed | 50
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- No Arms: All patient have a Quartet LV lead. No arms.
Arm/Group | No Arms
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Whose Cardiac Output (CO) Value in Acute, as Measured Echocardiographically, Improves With the Different Stimulation Vectors Offered by the Quartet® Left Ventricular Electrode.
Time Frame: Enrollment visit (in the seven days after implantation of the device)
Measure: Number; unit: participants
Arm/Group | No Arms
Number analyzed (Participants) | 51
participants | 27

2. Secondary Outcome: Percent Difference Between the Best CO From Non-traditional Vectors and Best CO From Traditional Vectors
Description: In patients with best CO obtained from Non-traditional, to calculate the percent difference between the best CO from Non-traditional vectors and best CO from Traditional vectors, vectors.This percentage was the CO from Non-traditional vectors minus CO from Traditional vectors then divided by CO from Traditional vectors.
  The Quartet® lead has 4 poles: Distal (D1), Mid 2 (M2), Mid 3 (M3) and Proximal (P4). The 3 Traditional vectors are the traditional configurations available in a standard bipolar lead: D1-M2, D1-Right Ventricular Coil (RVC) and M2-RVC. The 7 Non-traditional vectors are the additional configurations available in a Quartet® lead: D1-P4, M2-P4, M3-M2, M3-RVC, M3-P4, P4-M2 and P4-RVC.
Time Frame: At enrollment
Measure: Mean (Standard Deviation); unit: percentage of difference of CO
Arm/Group | No Arms
Number analyzed (Participants) | 51
percentage of difference of CO | 11.69 (11.12)

3. Secondary Outcome: Cardiac Output (CO) With Different Configurations at Enrollment
Description: Means of baseline non-paced CO, best CO obtained from traditional configurations and best CO obtained from all quadripolar configurations at enrollment.
Time Frame: Enrollment visit (in the seven days after implantation of the device)
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | No Arms
Number analyzed (Participants) | 51
L/min
  Non-paced CO | 3.64 (0.94)
  Best CO with Traditional vectors | 4.16 (1.12)
  Best CO with All vectors available in Quartet lead | 4.33 (1.12)

4. Secondary Outcome: Capture Threshold
Description: Capture and phrenic threshold data will be recorded for each of the stimulation vectors studied.
  Attempts will also be made to avoid phrenic stimulation in those patients who suffer from it, whilst maintaining good capture thresholds, by changing between the new configurations offered by the Quartet® electrode.
Time Frame: Enrollment visit (in the seven days after implantation of the device)
Measure: Mean (Standard Deviation); unit: volts
Arm/Group | No Arms
Number analyzed (Participants) | 51
volts
  Best Capture Threshold for Traditional vectors | 0.79 (0.47)
  Best Capture Threshold for Non-Traditional vectors | 0.97 (0.55)
  Best Capture Threshold for all vectors | 0.72 (0.32)

5. Secondary Outcome: Capture Threshold
Description: as for outcome 4
Time Frame: 6 months post-implant
Measure: Mean (Standard Deviation); unit: volts
Groups:
- Quartet LV Lead: All patient have a Quartet LV lead. No arms
Arm/Group | Quartet LV Lead
Number analyzed (Participants) | 50
volts
  Best Capture Threshold for Traditional vectors | 0.96 (0.54)
  Best Capture Threshold for Non-Traditional vectors | 1.21 (0.47)
  Best Capture Threshold for all vectors | 0.90 (0.41)

6. Secondary Outcome: Number of Vectors With Phrenic Nerve Stimulation (PNS)
Description: Capture and phrenic threshold data will be recorded for each of the stimulation vectors studied.
  Attempts will also be made to avoid phrenic stimulation in those patients who suffer from it, while maintaining good capture thresholds, by changing between the new configurations offered by the Quartet® electrode.
Time Frame: Enrollment visit (in the seven days after implantation of the device)
Measure: Number; unit: number of vectors
Units Other Than Participants: Number of total vectors
Arm/Group | No Arms
Number analyzed (Participants) | 51
Number analyzed (Number of total vectors) | 510
number of vectors
  Number of Traditional vectors with PNS | 51
  Number of Non-Traditional vectors with PNS | 69
  Number of Total vectors with PNS | 120

7. Secondary Outcome: Number of Vectors With Phrenic Nerve Stimulation (PNS)
Description: as for outcome 4
Time Frame: At 6 months
Measure: Number; unit: number of vectors
Units Other Than Participants: Number of vectors
Arm/Group | No Arms
Number analyzed (Participants) | 50
Number analyzed (Number of vectors) | 510
number of vectors
  Number of Traditional vectors with PNS | 49
  Number of Non-Traditional vectors with PNS | 69
  Number of Total vectors with PNS | 118

8. Secondary Outcome: Number of Patients With PNS in All Vectors
Description: To calculate the number of patients that exhibit PNS in all traditional vector
Time Frame: At enrollment
Measure: Number; unit: participants
Arm/Group | No Arms
Number analyzed (Participants) | 51
participants | 8

9. Secondary Outcome: Number of Patients With PNS in All Vectors, That Could be Avoided With a Non-traditional Vector
Description: To calculate the number of patients, who exhibit PNS in all traditional vector, in which PNS could be avoided using a non-traditional vector
Time Frame: At enrollment
Measure: Number; unit: participants
Arm/Group | No Arms
Number analyzed (Participants) | 51
participants | 7

10. Secondary Outcome: Number of Patients With PNS in All Vectors
Description: To calculate the number of patients that exhibit PNS in all traditional vector
Time Frame: At 6 months
Measure: Number; unit: participants
Arm/Group | No Arms
Number analyzed (Participants) | 50
participants | 7

11. Secondary Outcome: Number of Patients With PNS in All Vectors, That Could be Avoided With a Non-traditional Vector
Description: as for outcome 9
Time Frame: At 6 months
Measure: Number; unit: participants
Arm/Group | No Arms
Number analyzed (Participants) | 50
participants | 5

ADVERSE EVENTS:
Time Frame: 6 months period
Arm/Group | No Arms
Serious Adverse Events (participants affected / at risk) | 12/51
Other Adverse Events (participants affected / at risk) | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Arms (N=51)
RV lead dislodgment (Surgical and medical procedures) | 1 (1)
Dyspnea, angina pectoris, severe LV dysfunction, stent implantation (Cardiac disorders) | 1 (1)
Pneumothorax, lung was needled during implantation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
LV lead dislocation (Surgical and medical procedures) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Dyspnea due to renal failure, pulmonary edema, flutter (Cardiac disorders) | 1 (1)
Congestive cardiac insufficiency (Cardiac disorders) | 1 (1)
Renal insufficiency, cardiogenic shock and flutter (Cardiac disorders) | 1 (1)
Fever, infection (Infections and infestations) | 1 (1)
Fatigue, hypotension episode (Cardiac disorders) | 1 (1)
Atrial fibrillation, cardiovertion (Cardiac disorders) | 1 (1)
Dyspnea, acute lung edema after ICD explant and CRT implant Hypoxemia, COPD worsening renal failure (Cardiac disorders) | 1 (1)
Cognitive impairment, disorientation, injury from tumoral origin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal function worsening (Renal and urinary disorders) | 1 (1)
Pain at the pocket of device (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less